CLINICAL TRIAL: NCT05641285
Title: Diagnostic Utility of the Otosight Middle Ear Scope in Acute Otitis Media
Brief Title: Diagnostic Utility of Otosight Middle Ear Scope
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Anna Messner, Professor, Baylor College of Medicine
Other Study IDs: H-52641
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Ear Infection; Middle Ear Infection; Otitis Media
Keywords: Otoscope; Tympanogram
MeSH Terms: conditions — Otitis; Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Otosight, Otoscope, and Tympanogram: Prospective study using a convenience sample. There will be no group assignment or randomization. There is no intervention planned and therefore, no placebo group or use of controls.
  Interventions: Device: The OtoSight Middle Ear Scope

INTERVENTIONS:
Device: The OtoSight Middle Ear Scope — The OtoSight Middle Ear Scope is intended for use as an imaging tool for real-time visualization of the human tympanic membrane and fluid or air within the middle ear space. In the presence of middle ear fluid, the OtoSight Middle Ear Scope is used to visualize the fluid density. The OtoSight Middle Ear Scope is also used to provide surface images of the ear canal and tympanic membrane. It is indicated for use in children and adults.

SUMMARY:
Evaluate clinic workflow impact of OtoSight use for patients seen in the pediatric otolaryngology clinic.

DETAILED DESCRIPTION:
The purpose of this study is to compare the successful exam completion rate, the detection of middle ear fluid (versus no fluid), and the categorization of middle ear fluid (purulent vs. serous vs mucoid,) of routine otoscopy examination versus otosight examination versus tympanogram.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 months to 12 years old who are seen in the outpatient Otolaryngology clinic at Texas Children's Hospital main and west campuses.

Exclusion Criteria:

* Patients who have a history of ear tube placement

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged 6 months to 12 years old who are seen in the outpatient Otolaryngology clinic at Texas Children's Hospital main and west campuses who have no history of ear tube placement.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Exam Completion Rate | 6 months
  Compare the successful exam completion rate of these three diagnostic tools.
  For the Otosight device: presence or absence of visible tympanic membrane, and presence or absence of graph indicating fluid/no fluid in the middle ear.
  For tympanogram: presence or absence of interpretable tracing indicating normal tympanic membrane movement, retracted tympanic membrane, or no movement of tympanic membrane.
  For the Otoscope: success is visualization of the tympanic membrane versus unable to see tympanic membrane.
Detection of middle ear fluid | 6 months
  Compare the detection of middle ear fluid (versus no fluid) of these diagnostic tools.
Categorization of middle ear fluid | 6 months
  Compare the categorization of middle ear fluid (purulent vs. serous vs mucoid) of these diagnostic tools.

SECONDARY OUTCOMES:
Timed Evaluation of Clinic Flow | 6 months
  Evaluate clinic workflow impact of OtoSight use for patients seen in the pediatric otolaryngology clinic by timing how long it takes for the MA and/or MD to complete the Otosight exam.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Messner, MD, Principal Investigator — Baylor College of Medicine; Yi-Chun Liu, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No one besides the PI, the study staff, the IRB and the sponsor will have access to identifiable research data.